CLINICAL TRIAL: NCT06003569
Title: Reducing Asthma Attacks in Disadvantaged School Children With Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 20-0883; 5UG3HL151297 (NIH)
Record Dates: First submitted 2023-07-17; First posted 2023-08-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Asthma in Children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): School nurses/schools randomized to usual care will continue to receive their usual care from school nurses and then subsequently provide the intervention given their asthma remains poorly controlled at the start of the next school year following enrollment.
- BACK-S (Experimental): The BACK -Standard package includes a tailor-and-adapt to context strategy of approaches necessary to implement BACK in schools based on our past work, operationalized as an implementation blueprint to coordinate with partner roles of child/family, schools, healthcare teams and community resource agencies. This includes a facilitation strategy to support problem-solving through regular learning collaborative meetings for asthma navigators (bi-weekly), school nurses (monthly to bi-monthly) and health care champions (quarterly).
  Interventions: Behavioral: BACK-S
- BACK-E (Experimental): The BACK-Enhanced package includes the BACK-Standard package plus an Enhanced strategy to develop interrelationships with students/family, schools, and community agencies providing resources to address social determinants of health.
  Interventions: Behavioral: BACK-E

INTERVENTIONS:
Behavioral: BACK-S — BACK = Better Asthma Control for Kids:
  The BACK -Standard package includes a tailor-and-adapt to context strategy of approaches necessary to implement BACK in schools based on our past work, operationalized as an implementation blueprint to coordinate with partner roles of child/family, schools, healthcare teams and community resource agencies. This includes a facilitation strategy to support problem-solving through regular learning collaborative meetings for asthma navigators (bi-weekly), school nurses (monthly to bi-monthly) and health care champions (quarterly).
  Arms: BACK-S
Behavioral: BACK-E — The BACK-Enhanced package includes the BACK-Standard package plus an Enhanced strategy to develop interrelationships with students/family, schools, and community agencies providing resources to address social determinants of health.
  Arms: BACK-E

SUMMARY:
Our UH3 clinical trial, "Reducing Asthma Attacks in Disadvantaged School Children with Asthma," seeks broad-scale implementation of our effective school-based approach to improve asthma disparities for children, ages 5-12 years, in low-income communities. The investigators will contextualize dissemination and implementation (D&I) of our Colorado school-based asthma program (Col-SBAP) that reduces asthma exacerbations and missed school days, while also addressing social determinants of health. Our Better Asthma Control for Kids (BACK) Program will evaluate key metrics identified by diverse stakeholders during this dissemination trial in rural and small metropolitan areas of Colorado. Our clinical trial includes two implementation strategies: our standard Col-SBAP, titled BACK-Standard (BACK-S) and an enhanced community-centered approach, titled Back-Enhanced (BACK-E). These two strategies are designed for sustainable delivery by school asthma navigators and school nurses who coordinate with primary care and community resources. The Exploration, Preparation, Implementation, Sustainment (EPIS) D&I framework was applied with community partners during the UG3 planning phase to tailor implementation plans that meet local community needs, resources and priorities (EPIS Phases 1 & 2). BACK-S and BACK-E will be delivered from years 1-3 with data collection for implementation and effectiveness outcomes in 4 Colorado regions. In year 4, the investigators will collect data for sustainment outcomes (EPIS phase 3). The investigators will apply the work from EPIS phases 1-3 to refine our "dissemination playbook" that guides adoption by other school systems (EPIS Phase 4). Our primary implementation hypothesis is: Reach will be greater among students when delivered using the BACK-E arm as compared to BACK-S. Our effectiveness hypothesis is: BACK will be more effective than usual care at reducing asthma exacerbations. The BACK playbook includes training materials and a calculation of return on investment. The investigators are targeting schools with high levels of uncontrolled asthma and asthma associated burden. Our UH3 trial includes partner engagement to ensure BACK is disseminated to diverse geopolitical areas of Colorado with attention to sustainability. Collectively, our approach will accelerate dissemination of BACK nationally to communities experiencing health inequities in pediatric asthma care.

DETAILED DESCRIPTION:
Asthma disproportionately affects children living in disadvantaged communities. The well-documented disparities in asthma outcomes for minorities, including death, worse asthma control, greater likelihood of emergency room visits, and higher rates of school absenteeism are partly related to unmet SDOH for low-income families. Many SDOH contribute to uncontrolled asthma for low-income families, such as lack of insurance and transportation. For the child with asthma, this leads to reduced preventive care visits leading to more emergency visits and hospitalizations. Poor asthma control contributes to lower school performance due to missed school days and/fatigue and poorer concentration due to poor sleep quality. As a result, asthma is one of seven educationally relevant health disparities that school leaders seek to address to bend the widening achievement gap between low-income and higher income students. While some measures of health equity improved in the last decade, socio-economic disparities in asthma care have been stubbornly persistent.

A recent Cochrane review along with other reports identify key benefits of school-based asthma management programs, including reduced acute/urgent care health care use and days of restricted activity for students. Additionally, our work in this area for more than 15 years demonstrates improvements in self-management behaviors, quality of life, and school absenteeism. Core elements of our existing Colorado school-based asthma program (Col-SBAP) are concordant with those identified as effective in a Cochrane review, including education and counseling strategies to improve asthma knowledge and self-management skills to successfully control asthma. To date, these core Col-SBAP elements have been implemented in six school districts by school nurses and project funded asthma navigators (ANavs) - each ANav serves 40-65 children with uncontrolled asthma across one or more schools. A lesson learned during Col-SBAP implementation from our CABs is that the investigators need to address families' SDOH. Thus, the investigators developed a two-step intervention program, Col-SBAP combined with SDOH assessment/referral, termed Better Asthma Control for Kids (BACK). Our ANavs have had great success in identifying and addressing SDOH that directly impact asthma care, including inadequate insurance coverage, transportation, and difficulty affording medications. The core components of BACK are highly pragmatic and acceptable, as evidenced by the Denver Public School system sustaining Col-SBAP for 3 years with no external funding.

The investigators have developed, refined and piloted a program that is feasible to implement, and that has been sustained without external funding in one school district, but requires ongoing funding in other school districts. Support has largely come from public health agencies with limited engagement of Medicaid and other funders. To date, ours and others' work in school-based asthma care is also limited by the lack of generalizability to rural and smaller urban areas, and by the fact that our implementation guide does not help schools tailor implementation strategies to their community/site needs, resources, and priorities. Thus, the key next step to scale out BACK more broadly to use tools from the D&I field to prepare us for primetime dissemination and scalability. The UG3 award has allowed us to: 1) work purposively with multi-sectoral partners (including public health funders and insurers) in regions across Colorado where the investigators have not yet implemented our program to identify local needs, priorities and resources for BACK, and 2) tailor BACK implementation strategies to local factors. In the UH3 trial, the investigators will evaluate the effects of implementing BACK in diverse areas of Colorado, including rural regions with two different implementation packages, and will also identify different contextual factors that predict RE-AIM outcomes. Briefly, the investigators will identify how and why implementation strategies critical for local uptake and sustainability vary in their impact. Lessons learned will support the co-development of our BACK dissemination playbook with our partners so diverse and disadvantaged communities across the nation can feasibly implement BACK in a way that addresses local factors critical for success and sustainability.

Multi-sectoral engagement, including funders: The EPIS framework encourages the involvement of partners across multiple socioecological levels to support implementation. For BACK this includes patients/families, school health staff, primary care clinics, and community SDOH representatives that are part of our CABs. The investigators have also worked to engage health insurers and public health departments to ensure our implementation strategies consider payer perspectives and state public health integration.

Development Process for our Dissemination Playbook: The principles of "Designing for Dissemination" hold that it is critical to design evidence-based programs (EBPs) as a "product" that specifies not just core components, but details how to deliver the "product" within a site's usual way of practice. EPIS has been used previously to engage stakeholders to effectively package EBPs to tailor how implementation to address local needs and priorities. A key next step for future BACK dissemination is an innovative playbook to assist potential adopters to pick the types of "plays" needed to deliver the program with fidelity to core components but in a way that permits localized sustainability.

The investigators anticipate that typologies of context exist for each school site, such as the number of children eligible for BACK, needs and priorities for BACK, or the size of the school health team, that will influence implementation. Thus, the investigators propose to use our Aim 3a mixed methods evaluation to co-create a dissemination playbook prototype for implementation with our multi-sectoral partners, to help future adopters select implementation strategies tailored to their contextual typologies.

Innovative design of our playbook: Our dissemination playbook is innovative and extends the work of others by being interactive and allowing for site-specific tailoring through site self-evaluation assessments with immediate feedback identifying and suggesting relevant implementation strategies. It will permit tailoring to site to consider the general RE-AIM outcomes of BACK, including Reach to students and implementation costs. In addition, the playbook will allow school leaders to consider any significant variability of impact of BACK for different typologies of schools/communities (e.g., rural vs. urban, school nurse on-site yes/no). It will also highlight opportunities for reimbursement, including a bill to support community health worker reimbursement that was drafted by the Colorado House/Senate legislature in 2023.

Our specific aims for the UH3 trial phase are:

Aim 1: Among n=60 school nurses, their schools and students with poorly controlled asthma randomized to BACK-S vs. BACK-E in 4 regions of Colorado compare the reach (primary outcome), student retention, adoption, costs to future adopters, and sustainment.

Hypothesis 1a (Primary): Reach will be significantly greater among students with poorly controlled asthma when delivered using the BACK -E implementation package as compared to BACK-S package.

Aim 2: Determine and compare annual asthma exacerbation rates (i.e., exacerbations/year) in children with uncontrolled asthma randomized to either usual care (control) or the BACK intervention (using either the BACK-S or BACK-E implementation package).

Hypothesis 2: BACK will be more effective than usual care at reducing annual asthma exacerbations.

Aim 3a: Identify factors that predict student reach and retention, school-level adoption, costs to future adopters (schools), and sustainment for BACK-S or BACK-E.

Aim 3b: Based on the evaluation of Aims 1, 2 and 3a, adapt the current Denver based Col-SBAP, Asthma COMP implementation guide into a multi-media BACK dissemination playbook to guide the future dissemination of BACK (EPIS phase 4) Engagement of Multi-sectoral partners for Aims 1-3 Table 3 details the organization and membership in our partner groups. Drs. Szefler, Cicutto, Huebschmann, McFarlane and De Camp and Ms. Gleason formed community advisory boards (CAB) in 5 Colorado regions that met 3-4 times yearly in the UG3 phase and will continue to meet semi-annually in the UH3 phase. Our team will continue to work closely with the non-investigator elected chair to maintain engagement and effective group processes.

SCHOOL SITE RECRUITMENT:

Among the 5 school regions the investigators engaged with in the UG3 Phase, the investigators have successfully identified school nurses from four of the 5 regions for UH3 study participation. The 4 participating regions for the UH3 phase are the Lower Arkansas Valley (LAV), Delta/Mesa, Greeley/Weld/Fort Morgan, and Pikes Peak regions. The Montezuma/La Plata region was unable to engage with school districts to participate in the UH3 trial, but the investigators are maintaining the CAB in this region in anticipation of future BACK implementation.

School sites recruited serve socioeconomically diverse communities in rural and mid-size urban areas, representing ethnically/racially diverse populations that have SDOH characteristics placing them at higher risk of asthma burden. These include rural populations (e.g., the Lower Arkansas Valley, Morgan and Delta counties) and small-to-mid-size urban populations (e.g., Mesa County, Greeley), and large urban populations (Colorado Springs/Pikes Peak). The schools the investigators selected within each of the regions have >32% rates of free and reduced lunch, have a large proportion of minority children, and higher risk SDOH characteristics. The investigators will provide services in English and Spanish and employ bilingual ANavs.

APPROACH FOR AIMS 1-2 (UH3) Overarching objective: This research is guided by the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework and its emphasis on equity and representativeness. The investigators will study diverse and rural schools across four regions of Colorado and students with poor asthma control. In Aim 1, the investigators will compare reach and other implementation outcomes among schools and students with randomization at the school nurse level (n=~60) to deliver either the BACK-standard vs. BACK-enhanced implementation package. Separately, in Aim 2, the investigators will compare the effectiveness of the BACK intervention when delivered as either BACK-standard or BACK-enhanced, as compared to usual care. See Section 3D for specific aims.

PRAGMATIC UH3 STUDY DESIGN The investigators will conduct a pragmatic type 2 hybrid implementation-effectiveness trial; randomized at the level of school nurses, involving an open cohort, parallel cluster randomized trial where intervention conditions are phased in over two years. The investigators will compare the implementation outcomes of BACK-S and BACK-E with each other and will also compare the effectiveness outcomes (asthma exacerbations) of BACK-S/BACK-E with control arm.

ELIGIBILITY:
Inclusion Criteria:

* students with poor asthma control (or indicators of excess burden on school Asthma Intake Form)
* age 5-12 years of age
* attending one of participating schools in rural Colorado (school selection criteria: high rates of socioeconomic need based on high rates of free-and-reduced lunch or rural status)

Exclusion Criteria:

* age < 5 years or > 12 years
* students with no or controlled asthma

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Reach | Up to 48 months
  % of eligible students enrolled Numerator of Reach = number students consented with confirmed Asthma Intake Form (AIF) eligibility Denominator of Reach = number of eligible students
  o This denominator includes all students presumed eligible based on AIF at school registration, minus any students determined to NOT be eligible by AIF once the navigator called to confirm eligibility.

SECONDARY OUTCOMES:
Number of episode requiring systemic steroid therapy | Up to 48 months
  A reported number of episodes of systemic steroid therapy due to asthma, either orally or parenterally per year.
Number of ED/UC visits | Up to 48 months
  A reported number of Emergency Department (ED) and Urgent Care (UC) visits due to asthma per year.
Number of hospitalizations | Up to 48 months
  A reported number of hospitalizations due to asthma per year.

OTHER OUTCOMES:
Effectiveness based on asthma exacerbations | Up to 48 months
  Number of asthma exacerbations per year - defined as the number of asthma exacerbations requiring systemic steroid therapy, either orally or parenterally, following an ED visit, urgent care visit, hospitalization, or as directed by their clinician
Effectiveness based on missed school days | Up to 48 months
  Number of school days missed due to asthma per year
Adoption at a setting level | Up to 48 months
  % of eligible schools randomized to a study arm.
Planned Adoption at a staff level | Up to 48 months
  % of school nurses employed in an eligible school who agree to support the study intervention
Actual Adoption at a staff level | Up to 48 months
  % of school nurses employed in an eligible school who began supporting the study intervention
Fidelity to the intervention | Up to 48 months
  Fidelity to the intervention will be assessed as the percentage of participants that receive an adequate dose of the intervention, as defined by at least 2 of 3 planned intervention visits with students and at least 2 of 3 planned intervention visits with caregivers.
Implementation costs | Up to 48 months
  Total US dollar amount for the cost of the intervention materials and required resources
Maintenance | Up to 48 months
  Number of schools that continue to offer the intervention at 6-12 months after completion of active implementation support.
Sustainability | Up to 48 months
  Sustainability will be assessed in schools that have implemented the intervention with the Short Clinical Sustainability Assessment Tool (CSAT).
  * Minimum value: 1
  * Maximum value: 7
  * Interpretation guide: Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Amy G Huebschmann, MD, Principal Investigator — Childrens Hospital Colorado
Locations (13):
- United States (13):
  - Ault-Highland RE-9 school district, Ault, Colorado
  - Colorado Springs 11, Colorado Springs, Colorado
  - Harrison 2 school district, Colorado Springs, Colorado
  - Ellicott 22 school district, Ellicott, Colorado
  - Fountain 8 school district, Fountain, Colorado
  - Granada school district, Granada, Colorado
  - Greeley 6, Greeley, Colorado
  - East Otero R1 school district, La Junta, Colorado
  - Lamar RE2 school district, Lamar, Colorado
  - Las Animas school district, Las Animas, Colorado
  - Manzanola school district, Manzanola, Colorado
  - Weld County RE1, Platteville, Colorado
  - Wiggins RE-50(J), Wiggins, Colorado

IPD SHARING:
Plan to Share IPD: Yes
We will preserve and share all data generated in this project except data that cannot be shared safely because it is identifiable. We will put these data on the Open Science Framework (https://osf.io/) and embargo it. Additionally, during publication, we will make data available to share with reviewers.
Time Frame: August 2027
Access Criteria: Will be identified later

REFERENCES:
- [Background] Szefler SJ, Cicutto L, Brewer SE, Gleason M, McFarlane A, DeCamp LR, Brinton JT, Huebschmann AG. Applying dissemination and implementation research methods to translate a school-based asthma program. J Allergy Clin Immunol. 2022 Sep;150(3):535-548. doi: 10.1016/j.jaci.2022.04.029. Epub 2022 May 13. PMID 35569568
- [Background] Cicutto L, Gleason M, Haas-Howard C, White M, Hollenbach JP, Williams S, McGinn M, Villarreal M, Mitchell H, Cloutier MM, Vinick C, Langton C, Shocks DJ, Stempel DA, Szefler SJ. Building Bridges for Asthma Care Program: A School-Centered Program Connecting Schools, Families, and Community Health-Care Providers. J Sch Nurs. 2020 Jun;36(3):168-180. doi: 10.1177/1059840518805824. Epub 2018 Oct 18. PMID 30336726
- [Background] Cicutto L, Gleason M, Haas-Howard C, Jenkins-Nygren L, Labonde S, Patrick K. Competency-Based Framework and Continuing Education for Preparing a Skilled School Health Workforce for Asthma Care: The Colorado Experience. J Sch Nurs. 2017 Aug;33(4):277-284. doi: 10.1177/1059840516675931. Epub 2016 Nov 30. PMID 28726584
- [Background] Waltz TJ, Powell BJ, Fernandez ME, Abadie B, Damschroder LJ. Choosing implementation strategies to address contextual barriers: diversity in recommendations and future directions. Implement Sci. 2019 Apr 29;14(1):42. doi: 10.1186/s13012-019-0892-4. PMID 31036028
- [Background] Kneale D, Harris K, McDonald VM, Thomas J, Grigg J. Effectiveness of school-based self-management interventions for asthma among children and adolescents: findings from a Cochrane systematic review and meta-analysis. Thorax. 2019 May;74(5):432-438. doi: 10.1136/thoraxjnl-2018-211909. Epub 2019 Jan 27. PMID 30686788
- [Background] Walter H, Sadeque-Iqbal F, Ulysse R, Castillo D, Fitzpatrick A, Singleton J. Effectiveness of school-based family asthma educational programs in quality of life and asthma exacerbations in asthmatic children aged five to 18: a systematic review. JBI Database System Rev Implement Rep. 2016 Nov;14(11):113-138. doi: 10.11124/JBISRIR-2016-003181. PMID 27941517
- [Background] Akinbami LJ, Moorman JE, Simon AE, Schoendorf KC. Trends in racial disparities for asthma outcomes among children 0 to 17 years, 2001-2010. J Allergy Clin Immunol. 2014 Sep;134(3):547-553.e5. doi: 10.1016/j.jaci.2014.05.037. Epub 2014 Aug 1. PMID 25091437
- [Background] Cicutto L, Murphy S, Coutts D, O'Rourke J, Lang G, Chapman C, Coates P. Breaking the access barrier: evaluating an asthma center's efforts to provide education to children with asthma in schools. Chest. 2005 Oct;128(4):1928-35. doi: 10.1378/chest.128.4.1928. PMID 16236837
- [Background] Cicutto L, To T, Murphy S. A randomized controlled trial of a public health nurse-delivered asthma program to elementary schools. J Sch Health. 2013 Dec;83(12):876-84. doi: 10.1111/josh.12106. PMID 24261522
- [Background] Szefler SJ, Cloutier MM, Villarreal M, Hollenbach JP, Gleason M, Haas-Howard C, Vinick C, Calatroni A, Cicutto L, White M, Williams S, McGinn M, Langton C, Shocks D, Mitchell H, Stempel DA. Building Bridges for Asthma Care: Reducing school absence for inner-city children with health disparities. J Allergy Clin Immunol. 2019 Feb;143(2):746-754.e2. doi: 10.1016/j.jaci.2018.05.041. Epub 2018 Jul 25. PMID 30055181
- [Background] Cicutto L, To T, Murphy S. Cicutto, To, and Murphy respond: a randomized controlled trial of a public health nurse-delivered asthma program to elementary schools. J Sch Health. 2014 Jun;84(6):350. doi: 10.1111/josh.12163. No abstract available. PMID 24749915
- [Background] Liptzin DR, Gleason MC, Cicutto LC, Cleveland CL, Shocks DJ, White MK, Faino AV, Szefler SJ. Developing, Implementing, and Evaluating a School-Centered Asthma Program: Step-Up Asthma Program. J Allergy Clin Immunol Pract. 2016 Sep-Oct;4(5):972-979.e1. doi: 10.1016/j.jaip.2016.04.016. Epub 2016 Jun 7. PMID 27283054
- [Background] Feldstein AC, Glasgow RE. A practical, robust implementation and sustainability model (PRISM) for integrating research findings into practice. Jt Comm J Qual Patient Saf. 2008 Apr;34(4):228-43. doi: 10.1016/s1553-7250(08)34030-6. PMID 18468362
- [Background] Gleason M, Cicutto L, Haas-Howard C, Raleigh BM, Szefler SJ. Leveraging Partnerships: Families, Schools, and Providers Working Together to Improve Asthma Management. Curr Allergy Asthma Rep. 2016 Oct;16(10):74. doi: 10.1007/s11882-016-0655-0. PMID 27709456
- [Background] Powell BJ, Waltz TJ, Chinman MJ, Damschroder LJ, Smith JL, Matthieu MM, Proctor EK, Kirchner JE. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. Implement Sci. 2015 Feb 12;10:21. doi: 10.1186/s13012-015-0209-1. PMID 25889199
- [Background] Waltz TJ, Powell BJ, Matthieu MM, Damschroder LJ, Chinman MJ, Smith JL, Proctor EK, Kirchner JE. Use of concept mapping to characterize relationships among implementation strategies and assess their feasibility and importance: results from the Expert Recommendations for Implementing Change (ERIC) study. Implement Sci. 2015 Aug 7;10:109. doi: 10.1186/s13012-015-0295-0. PMID 26249843
- [Background] Proctor EK, Powell BJ, McMillen JC. Implementation strategies: recommendations for specifying and reporting. Implement Sci. 2013 Dec 1;8:139. doi: 10.1186/1748-5908-8-139. PMID 24289295
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] Glasgow RE, Estabrooks PE. Pragmatic Applications of RE-AIM for Health Care Initiatives in Community and Clinical Settings. Prev Chronic Dis. 2018 Jan 4;15:E02. doi: 10.5888/pcd15.170271. PMID 29300695
- [Background] Malone S, Prewitt K, Hackett R, Lin JC, McKay V, Walsh-Bailey C, Luke DA. The Clinical Sustainability Assessment Tool: measuring organizational capacity to promote sustainability in healthcare. Implement Sci Commun. 2021 Jul 17;2(1):77. doi: 10.1186/s43058-021-00181-2. PMID 34274004
- [Derived] Huebschmann AG, Wagner NM, Gleason M, Brinton JT, Brtnikova M, Brewer SE, Begum A, Armstrong R, DeCamp LR, McFarlane A, DeKeyser H, Coleman H, Federico MJ, Szefler SJ, Cicutto LC. Reducing asthma attacks in disadvantaged school children with asthma: study protocol for a type 2 hybrid implementation-effectiveness trial (Better Asthma Control for Kids, BACK). Implement Sci. 2024 Aug 15;19(1):60. doi: 10.1186/s13012-024-01387-3. PMID 39148094
- See also: SDOH determination — https://health.gov/healthypeople/priority-areas/social-determinants-health
- See also: Consolidated Framework for Implementation Research - Implementation Strategy Matching Tool — https://cfirguide.org/choosing-strategies/
- See also: Public school students eligible for free or reduced-price lunch — https://nces.ed.gov/FastFacts/display.asp?id=898

DOCUMENTS (1):
  • Informed Consent Form (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT06003569/ICF_000.pdf